CLINICAL TRIAL: NCT04342637
Title: Gastrointestinal Endoscopy in the Era of COVID-19: a Multinational Survey
Brief Title: COVID-19 Endoscopy Survey
Acronym: COVID-19 Endo
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Lecturer of medicine and gastroenterology, Al-Azhar University
Other Study IDs: WES-2
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: Endoscopy; Gastrointestinal; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Practicing gastroenterologists: Practicing physicians performing gastrointestinal endoscpy
  Interventions: Other: Practice details

INTERVENTIONS:
Other: Practice details — Physicians will report details of their endoscopy practice through answering the questions of the questionnaire

SUMMARY:
A questionnaire containing some critical questions about practice inside GI endoscopy units in different countries will be distributed via emails. Responses will be collected in an online platform and data will be analyzed to reveal the effect of SARS-CoV-2 pandemic on different aspects of GI endoscopy practice in the studied countries.

DETAILED DESCRIPTION:
Participants has to answer the following questions:

1. Participating center data:

   * Participant name (surname, first name): (optional)
   * Participant email: (optional)
   * Country: ……..
   * Working days (before COVID-19): ……..
   * Types of procedure performed /day (before COVID-19): …….
   * Number of endoscopists /day (before COVID-19): …….
   * Number of nursing staff /day (before COVID-19): …….
   * Number of administrative staff /day (before COVID-19): …….
   * Number of patients undergoing endoscopy/ day (before COVID-19): …….
   * Availability of negative pressure rooms (before COVID-19): …….
   * Number of endoscopy referrals/ day (before COVID-19): ……..
2. Response to COVID-19:

   * Working days (after COVID-19): ……..
   * Types of procedure performed /day (after COVID-19): ……..
   * Number of endoscopists /day (after COVID-19): ……..
   * Number of nursing staff /day (after COVID-19): ……..
   * Number of administrative staff /day (after COVID-19): ……..
   * Do you consider teams (MD, RN, tech, anesthesia) that remain together for the entire day so as to compartmentalize and minimize personnel exposure?
   * Number of patients undergoing endoscopy/ day (after COVID-19): ……..
   * Number of endoscopy referrals/ day (after COVID-19): ……..
   * Availability of negative pressure rooms or use portable industrial-grade high-efficiency particulate air (HEPA) filters as a reasonable alternative: ……..
   * Which recommendations do you follow? WEO, AGA, BSG, APSDE, other
   * Applying triage for patients: e.g. FTOCC (APSDE); dose this include any tests
   * Do you use any of this for triage of patients: i) a telephone consultation with the referring provider or (ii) a telehealth visit with the patient or (iii) a multidisciplinary team approach or (virtual) disease/tumor board to facilitate decision-making for complicated patients.
   * Prioritization:

Which classification do you use for endoscopic procedures?

1. urgent, semi-urgent and elective during COVID-19 outbreak
2. Time sensitive procedure:

   * Time-sensitive procedures defined as procedures that if deferred may negatively impact patient-important outcomes. The decision to defer a procedure should be made on a case-by-case basis:
   * Time-Sensitive* (within 24 hours-8 weeks):

     1. Threat to the patient's life or Permanent dysfunction of an organ e.g. diagnosis and treatment of GI bleeding or cholangitis
     2. Risk of metastasis or progression of stage of disease e.g. e.g. work up of symptoms suggestive of cancer
     3. Risk of rapidly worsening progression of disease or severity of symptoms e.g. management decisions, such as treatment for IBD
   * Non-Time Sensitive: No short-term impact on patient-important outcomes e.g. screening or surveillance colonoscopy, follow up colonoscopy for +FIT
   * What are the most common clinical presentations? (please choose all that apply): Upper GI bleeding, lower GI bleeding, cholangitis, suspected cancer, foreign body, relive of GI obstruction, gastrostomy, other
3. Endoscopy and use of PPE:

   * Did you receive appropriate education and training on infection control measures, including hand hygiene.
   * Did you receive adequate training on gowning and removal of PPE?
   * Do you practice Standard hand hygiene procedures before and after each case?
   * What type of personal protective equipment (PPE) do you usually use for doing an endoscopic procedure nowadays? (choose all that apply)

   Surgical mask N95 mask Isolation gown with water resistance Head cover Eye protection Face shield N95 protection in combination with face shield or surgical mask Other (please specify): ……..
   * Do you extend (over 8 hours) use of N95 masks?
   * Do you re-use of N95 masks?
   * Do you extend use (over 8 hours) any other equipment? : …..
   * Do you re use any other equipment? …..
   * If yes, please specify: …… If yes please specify: …..
   * Do you use of double gloves? ……
   * What PPE do you use for the following cases (choose all that apply)?

     1. Suspected cases of SARS-CoV-2 infection:

        Surgical mask N95 mask isolation gown with water resistance head cover eye protection face shield negative pressure room other please specify
     2. Probable cases of SARS-CoV-2 infection:

        Surgical mask N95 mask isolation gown with water resistance head cover eye protection face shield negative pressure room other please specify
     3. confirmed cases of SARS-CoV-2 infection: Surgical mask N95 mask isolation gown with water resistance head cover eye protection face shield negative pressure room other please specify
4. Post endoscopy:

   * Do you motion in your report the status of the patients (suspected, probable, confirmed case of SARS-CoV-2 infection?
   * Do you use standard endoscopic decontamination or anything extra?
   * Do you give time for sterilizing endoscopy room after each suspected or confirmed case of SARS-CoV-2 infection? How long?
   * Do you call back your patients 2 weeks after procedure to ask them about symptoms/ diagnosis of SARS-CoV-2 infection?
   * Did you report any endoscopy related SARS-CoV-2 infection in your center (anytime for HCWs & up to two weeks after procedures for patients)?
   * Are you preparing a management plan for the waiting list after the current phase of the pandemic?

ELIGIBILITY:
Inclusion Criteria:

* physicians working in endoscopy units worldwide

Exclusion Criteria:

* physicians not working in endoscopy units worldwide

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - physicians working and practicing in gastrointestinal endoscopy units worldwide
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of GI societies recommendations on prevention of SARS-CoV-2 infection | 4- 6 months
  To evaluate the validity of different GI societies recommendations applied locally and how effective they are in preventing transmission in endoscopy units through reporting any new cases developing COVID-19 within two weeks of doing endoscopy (whether a patient or health-care worker)
To measure the percentage change in performed endoscopic procedure in response to COVID-19 | 4- 6 months
  To measure the percentage change in performed endoscopic procedure in response to COVID-19 in different centers of the world and the alternative solutions given to overcome this problem.

SECONDARY OUTCOMES:
Effect of COVID-19 precautions on procedure time | 4- 6 months
  Effect of COVID-19 precautions on procedure time
Effect of COVID-19 precautions on time of disinfection | 4- 6 months
  Effect of COVID-19 precautions on prolongatIon of time of disinfection
Effect of COVID-19 precautions on procedure success | 4- 6 months
  Effect of COVID-19 precautions on the ability of the endoscopist to finish the procedure successfully
Effect of COVID-19 precautions on complications | 4- 6 months
  Effect of COVID-19 precautions on occurrence of complications
Effect of COVID-19 precautions on working time | 4- 6 months
  Effect of COVID-19 precautions on change of working time (prolongation or shortening)
Effect of COVID-19 precautions on staff number | 4- 6 months
  Effect of COVID-19 precautions on change of staff number

CONTACTS AND LOCATIONS:
Locations (4):
- Kings County Hospital Center, Brooklyn, NY, USA, Albertson, New York, United States
- Egypt (2):
  - Faculty of Medicine, Zagazig University, Zagazig, Sharqia Province
  - Al-Azhar Univerisity, Cairo
- Ahvaz Imam hospital, Ahvāz, Iran

IPD SHARING:
Plan to Share IPD: Undecided
After publication we may share data

REFERENCES:
- [Result] Ruuskanen O, Lahti E, Jennings LC, Murdoch DR. Viral pneumonia. Lancet. 2011 Apr 9;377(9773):1264-75. doi: 10.1016/S0140-6736(10)61459-6. Epub 2011 Mar 22. PMID 21435708
- [Result] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Result] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Result] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Result] Sultan S, Lim JK, Altayar O, Davitkov P, Feuerstein JD, Siddique SM, Falck-Ytter Y, El-Serag HB; AGA Institute. Electronic address: ewilson@gastro.org. AGA Rapid Recommendations for Gastrointestinal Procedures During the COVID-19 Pandemic. Gastroenterology. 2020 Aug;159(2):739-758.e4. doi: 10.1053/j.gastro.2020.03.072. Epub 2020 Apr 1. No abstract available. PMID 32247018
- [Result] Chiu PWY, Ng SC, Inoue H, Reddy DN, Ling Hu E, Cho JY, Ho LK, Hewett DG, Chiu HM, Rerknimitr R, Wang HP, Ho SH, Seo DW, Goh KL, Tajiri H, Kitano S, Chan FKL. Practice of endoscopy during COVID-19 pandemic: position statements of the Asian Pacific Society for Digestive Endoscopy (APSDE-COVID statements). Gut. 2020 Jun;69(6):991-996. doi: 10.1136/gutjnl-2020-321185. Epub 2020 Apr 2. PMID 32241897
- See also: WHO: Coronavirus Disease 2019 (COVID-19): Situation Report--51. WHO website. Published March 11, 2020. Accessed April 6, 2020. — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200311-sitrep-51-covid-19.pdf
- See also: WEO COVID-19 Response Taskforce. WEO Advice to Endoscopists. accessed April 7, 2020. — https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf